CLINICAL TRIAL: NCT01803945
Title: A Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AVE8112 in Patients With Parkinson's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: First milestone was not met.
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MJFF AVE8112 MAD PD
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; cognitive impairment; movement disorder
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Group (Placebo Comparator): Sequential cohorts of eight patients with PD will be administered ascending oral doses of AVE8112 (n=6) or placebo (n=2) once a day for 14 days. Patients will be assessed in clinic for 30 hours following the initial oral dose of AVE8112 or placebo
  Interventions: Drug: Placebo
- AVE8112 (Active Comparator): Sequential cohorts of eight patients with PD will be administered ascending oral doses of AVE8112 (n=6) or placebo (n=2) once a day for 14 days. Dosing for subsequent cohorts will only proceed, and the dose level selected, after the safety and tolerability of the previous cohort has been reviewed. Doses are planned to be 1.0, 2.0, 3.0, and 4.0 mg once a day for 14 days. These are planned treatments, but doses may be modified based on safety review of previous cohort(s). In addition, cohorts may be added to reconfirm a previously administered dose, and/or a titration strategy may be employed to reach a desired dose. Patients will be assessed in clinic for 30 hours following the initial oral dose of AVE8112 or placebo
  Interventions: Drug: AVE8112

INTERVENTIONS:
Drug: AVE8112
  Arms: AVE8112
Drug: Placebo
  Arms: Placebo Group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple-ascending dose study of orally administered AVE8112 in patients with Parkinson's Disease (PD).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multiple-ascending dose study of orally administered AVE8112 in patients with Parkinson's Disease (PD). Sequential cohorts of eight patients with PD will be administered ascending oral doses of AVE8112 (n=6) or placebo (n=2) once a day for 14 days. Dosing for subsequent cohorts will only proceed, and the dose level selected, after the safety and tolerability of the previous cohort has been reviewed. Doses are planned to be 1.0, 2.0, 3.0, and 4.0 mg once a day for 14 days. These are planned treatments, but doses may be modified based on safety review of previous cohort(s). In addition, cohorts may be added to reconfirm a previously administered dose, and/or a titration strategy may be employed to reach a desired dose.

Patients will be assessed in clinic for 30 hours following the initial oral dose of AVE8112 or placebo. Subsequent dosing will occur on an outpatient basis. Patients will receive telephone calls on Days 3 and 10 to monitor for adverse events (AEs) and concomitant medications, and will also be assessed in the clinic on Study Days 7 (outpatient), 14 (outpatient), and 28 (± 3 days) (Follow-up visit). Safety assessments will include physical examinations, vital signs, ECGs, clinical laboratory evaluations, Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS), and Columbia Suicide Severity Rating Scale (C-SSRS). Pharmacodynamic assessment will include the Parkinson's Disease Cognitive Rating Scale (PD-CRS).

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 to 70, inclusive, with a diagnosis of PD, currently being treated with a stable regimen (at least 4 weeks) of anti-parkinsonian drugs which include at least one L 3,4 dihydroxyphenylalanine (L DOPA)-containing therapy with or without dopamine agonist at Screening.
* Patients must have at least two of the following: resting tremor, bradykinesia, rigidity (must have either resting tremor or bradykinesia), or gait disturbances as assessed during physical/neurological exam at the Screening visit.
* A diagnosis of PD for 10 years or less at Screening.
* Hoehn and Yahr stage I - III.
* Male or female age 30 years or older at time of PD diagnosis.
* Body Mass Index (BMI) of approximately ≥18 to ≤32 kg/m2; and a total body weight > 50 kg (l10 lbs).
* Female patients must be of non-childbearing potential.

Exclusion Criteria:

* Clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s) as determined by the Investigator or designee.
* Female patients that are breastfeeding or female patients with a positive serum pregnancy test.
* Use of cholinergic medications or those with cholinergic effects.
* History of orthostatic hypotension or symptomatic drop in SBP.
* Any subject who has advanced Parkinson's Disease.
* Evidence of severe depression (score of >10 on Quick Inventory of Depressive Symptomatology - Self Rated [QIDS-SR]).
* Personal and/or familial history of a significant suicide attempt.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Continuous; Patients will be assessed for a period of 28 days

SECONDARY OUTCOMES:
Pharmacodynamics | Continuous; Patients will be assesed for a period of 28 days
Pharmacokinetics | Continuous; Patients will be assessed for a period of 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - California Clinical Trials, Glendale, California
  - PARAXEL International, Baltimore, Maryland